CLINICAL TRIAL: NCT05073757
Title: Prospective Study to Evaluate the Performance and Safety of Personalized Implants in Cranio-Maxillofacial (CMF) Surgery Indicated for Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: Global D (Industry)
Responsible Party: Sponsor
Other Study IDs: 2001-S-CMF-SUR MESURE-R
Record Dates: First submitted 2021-08-04; First posted 2021-10-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Surgery; Orthognathic Surgery; Orthognathic Surgical Procedures
Keywords: orthognatic surgery; guided surgery; 3D printing; plate; screw; custom-made
MeSH Terms: interventions — Bone Plates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthognatic surgery: Orthognathic surgery patients, adults or minors whose bone maturity is sufficient according to the investigator.
  Interventions: Device: Custom-made guides and plates

INTERVENTIONS:
Device: Custom-made guides and plates — Patients will be included in the study and then followed clinically according to the routine care of orthognathic surgery with custom-made guides and plates. The only specific act of this study is the completion of an OQLQ quality of life questionnaire by patients preoperatively and between 8 to 12 months postoperatively.

SUMMARY:
With the digital age, guided surgery and cases of fully computer-assisted surgeries via 3D printing guides and preformed plates are booming.

Our project aims to study the performance and safety of custom-made implants (custom-made guides and plates) in orthognathic surgery in order to obtain specific clinical data on SLS France devices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, adult or minor having reached bone maturity according to the judgment of the investigator,
* Patient having first orthognathic surgery with SLS France custom-made guides and plates,
* Patient who received orthodontic treatment prior to orthognathic surgery,
* Patient able to read, understand and answer the study quality of life questionnaire,
* Patient (and legal representative if a minor) who is not opposed to his participation in the study or to the processing of his data.
* Patient affiliated to a social insurance

Exclusion Criteria:

* Patient allergic to one of the compounds of the plates and / or guides,
* Patient with physical or mental disability making it impossible to follow up in the study,
* Patient with significant expansion
* Patient with a congenital craniofacial malformation
* Patient with acute or chronic local or systemic infection,
* Person placed under legal protection,
* Pregnant or breastfeeding women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Orthognatic surgery male or female patients, adults or minors whose bone maturity is sufficient according to the judgment of the investigator.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Orthognatic quality of life questionnaire | 12 months post-operatively
  To evaluate the performance of custom-made implants indicated for orthognathic surgery by measuring the quality of life of patients

SECONDARY OUTCOMES:
Surgeon satisfaction on the implant's utilisation | Immediately following surgery
  Assessment by a satisfaction questionnaire, specially developed for the study, completed by the surgeon after the surgery. The surgeon evaluates each item using a likert scale (Highly Satisfied/ Satisfied/ Not very satisfied / Unsatisfied).
Security of the implants used for orthognathic surgery | 12 months
  Adverse events identification, assessment and follow-up.

CONTACTS AND LOCATIONS:
Locations (4):
- Cabinet chirurgie Maxillo-faciale, Tournai, Belgium
- France (3):
  - Cabinet Orhognatic, Lyon
  - Hôpital de la Loire, Saint-Etienne
  - Hôpital Villefranche sur Sâone, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No